CLINICAL TRIAL: NCT06837285
Title: Real-World Assessment of Clinical Evidence for Mandibular Advancement Treatment of Obstructive Sleep Apnea
Brief Title: Clinial Study of Treatment With Mandibular Advancement Device in Patients With Obstructive Sleep Apnea Across 6 General Hospitals
Acronym: RACEMADT
Status: Completed | Type: Observational
Sponsor: University Hospital, Antwerp (Other)
Collaborators: AZ Sint-Maarten (Unknown); AZ Voorkempen (Unknown); AZ Monica Campus Antwerpen (Unknown); Imelda Hospital, Bonheiden (Other); Vitaz (Other); Heilig Hart Ziekenhuis Lier (Unknown)
Responsible Party: Principal Investigator, Marc Braem, em. prof. dr., University Hospital, Antwerp
Other Study IDs: EVO_AZ-Sites_2025
Record Dates: First submitted 2025-02-10; First posted 2025-02-20 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Obstructive Sleep Apnea (OSA); Mandibular Advancement Device
Keywords: obstructive sleep apnea; non invasive therapy; mandibular advancement device
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Occlusal Splints

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

INTERVENTIONS:
Device: mandibular advancement device — Results of clinical trials on MADs are regularly published in the international literature but are generally very strongly controlled studies, still far away from being applied in routine daily clinical practice. The current retrospective study evaluates real-world data to determine the extent to which MAD improves both symptoms in patients with OSA. It is estimated that about 3% of newly diagnosed OSA patients are treated with MAD. In the light of new future treatment conventions, health government departments are increasingly demanding real-world data to stimulate knowledge of the relative effectiveness and value of treatments in the management of patients in routine clinical settings.

SUMMARY:
Study Objectives: To retrospectively study mandibular advancement treatment efficacy using apnea-hypopnea index (AHI) and oxygen desaturation index (ODI), in a large cohort of patients, in 'real world' settings across 6 general hospitals.

Methods: Diagnosis at 6 Belgian recognised OSA sleepcenters with type-1 polysomnography. After drug-induced sleep endoscopy by Ear-Nose-Troat-specialist, patients with positive effect of mandibular protrusion on reopening the upper airway were referred. The mandibular advancement device (MAD) was fitted in 'maximal comfortable protrusion' minus 2mm. A type-3 home polygraphy with MAD followed titration.

DETAILED DESCRIPTION:
Methods Patients were diagnosed at conventionalized Belgian OSA sleep centers, in alphabetical order: AZ Monica (Antwerpen), AZ Sint-Maarten (Mechelen), AZ Voorkempen (Malle), Heilig Hart Ziekenhuis (Lier), Imelda Ziekenhuis (Bonheiden), and VITAZ (Sint-Niklaas), with a type 1 polysomnography. The apnea-hypopnea index (AHI; number of events/h sleep), oxygen desaturation index (ODI; number of desaturations/h sleep) and body mass index (BMI; kg/m2) were calculated.

The Ear-Nose-Troat-specialist at the OSA sleep center performed an awake examination of the upper airway, followed by a drug-induced sleep endoscopy (DISE). Patients with positive effect of mandibular protrusion on reopening of the upper airway were referred to the dental sleep professional (DSP) for dental clinical and/or radiological examination. The DSP registered the mandibular protrusive trajectory with a bite registration device (The BiteFix, Scheu-Dental, Iserlohn, Germany) and a hard bite registration paste (Futar Fast, Kettenbach, Germany), as to achieve a stable fit on both tooth arcs. Next, the 'maximal comfortable protrusion' (MCP, mm) of the mandible was determined, being the most forward mandibular protrusion still tolerated by the patient and tested during DISE.

At the time of fitting, the patients received full explanation on the MAD titration schedule and were instructed to titrate after fitting of the MAD till resolution of the snoring symptoms or upon reaching physiological limits. A 1-month follow-up was performed by telephone. Next, a type 3 home polygraphy with the MAD was organized between 3 to 5 months after treatment start, recording identical parameters as at baseline, making each patient to serve as the own control.

Inclusion In Belgium, the reimbursement criterion for MADt leaves out central apneas in the calculation of AHI and requires this 'obstructive AHI' (OAHI) to be ≥ 15 events/h. In the absence of any central event, the OAHI = AHI, whereas in the presence of central events OAHI < AHI. Patients with OAHI ≥ 15 events/h and therefore AHI ≥ 15 events/h were included on the condition that the full clinical pathway as described before was followed and that the MAD was self-reportedly used at least 4 hours per night. Further reporting is done on AHI, for reasons of comparison with other studies.

Parameters Age (years) and gender (Male/Female, M/F) were noted. Questionnaires were used at baseline and controls for the quantification of snoring using a visual analogue score on loudness (VAS-snore) with a Likert-scale from 0 (no snoring) up to 10 (partner sleeps in other room). A VAS-snore > 3/10 represents socially disturbing snoring. The Epworth sleepiness score (ESS) quantifies daytime sleepiness with ESS ≥ 11/24 representing increased propensity to fall asleep during daytime.

Mandibular advancement device The starting position of the MADt was set at MCP minus 2mm (MCP-2, mm). Digital imprints of both tooth arcs were taken (Trios, 3Shape, Copenhagen, Denmark) as well of the bite-registration in the MCP-2 position. The selected MAD (EVO, ProSomnus Sleep Technologies, Pleasanton, CA, USA) uses a Class IV resin (United States Pharmacopeia and National Formulary) which is the highest grade of material currently available. Its design is characterized by perpendicular rectangular posts to protrude the mandible. Such design could preserve mandibular advancement even during limited mouth opening while asleep. The fully digital manufacturing pathway, starting from the digital intra-oral scans up to the 3D milling, favors accuracy-of-fit on the dental arcs.

ELIGIBILITY:
Inclusion Criteria:

* obstructive apnea-hypopnea index ≥ 15 events/h sleep
* complete clinical pathway

Exclusion Criteria:

* obstructive apnea-hypopnea index < 15 events/h sleep
* not dental fit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients referred by sleep physicians and after ear-nos-troat-specialist examination, for mandibular advancement treatment in routine clinical settings.
Sampling Method: Probability Sample
Enrollment: 182 (Actual)
Dates: Start 2021-09-22 (Actual); Primary Completion 2024-10-24 (Actual); Study Completion 2024-10-24 (Actual)

PRIMARY OUTCOMES:
Respiratory index "apnea-hypopnea index" (AHI) | From enrollment to the control home polygraphy at 3 to 5 months after fitting the MAD
  The first primary outcome is an expected improvement in apnea-hypopnea index (AHI; number of apneas and hypopneas per hour of sleep; a higher AHI means more severe obstructive sleep apnea) upon MAD treatment (MADt). Functional objective outcome measure is the quantification of the effect of MADt on AHI. "Success" is defined as treatment AHI≤15 events/h following the Belgian threshold for reimbursement, and any decrease in baseline AHI.
Respiratory index "oxygen desaturation index" (ODI) | From enrollment to the control home polygraphy at 3 to 5 months after fitting the MAD
  The second primary outcome is an expected improvement in respiratory parameter oxygen desaturation index (ODI; number of desaturations per hour of sleep; a higher ODI means a more severe condition) upon MAD treatment (MADt). Functional objective outcome measure is the quantification of the effect of MADt on ODI. "Success" is defined as treatment AHI≤15 events/h following the Belgian threshold for reimbursement, and any decrease in baseline AHI.
Obstructive sleep apnea severity | From enrollment to the control home polygraphy at 3 to 5 months after fitting the MAD
  The third primary outcome is an expected improvement in OSA severity category upon MAD treatment (MADt). Categories are defined as AHI 5-14.9/hour = mild OSA; AHI 15-29.9/hour = moderate OSA; and OSA ≥30/hour = severe OSA.
Visual analogue score for snoring | From enrollment to the control home polygraphy at 3 to 5 months after fitting the MAD
  The fourth primary outcome is an expected improvement in snoring as reported by the patient. This functional subjective outcome measure quantifies the snoring using a questionnaire with a visual analogue score on loudness of snoring (VAS-snore) with a Likert-scale from 0 (no snoring) up to 10 (partner sleeps in other room). A VAS-snore > 3/10 represents socially disturbing snoring. The higher the VAS-snore score the louder the snoring is.
Epworth Sleepiness Scale | From enrollment to the control home polygraphy at 3 to 5 months after fitting the MAD
  The fifth primary outcome is an expected improvement in daytime sleepiness as reported by the patient. This functional subjective outcome measure quantifies the propensity to fall asleep during daytime activities, using a questionnaire with with the Epworth Sleepiness Score-scale (ESS) from 0 (no propensity to fall asleep) up to 24 (extremely high propensity to fall asleep). An EES-score ≥ 11/24 represents a pathological increased daytime sleepiness. The higher the ESS-score the more pronounce the daytime sleepiness is.
Titration | From enrollment to the control home polygraphy at 3 to 5 months after fitting the MAD
  The sixth primary outcome is the amount of titration required at the moment when the control home-polygraphy (HPG) is recorded. The starting position of the MADt was set at the maximal comfortable protrusion (MCP) minus 2mm: first the mandibular maximal protrusive trajectory was measured in millimeters. Next, MCP was determined, being the most forward mandibular protrusion still tolerated by the patient. The actual protrusive position of the MAD at the time of the HPG minus the start position quantifies the amount of protrusion. This result cannot be interpreted in terms of a 'higher' protrusion as a 'better' protrusion since this is a patient specific characteristic, as is the range of mandibular protrusion.

CONTACTS AND LOCATIONS:
Overall Officials: Marc J BRAEM, DDS, PhD, Principal Investigator — UZA Afd. Tandheelkunde
Locations (6):
- Belgium (6):
  - AZ Voorkempen, Malle, Antwerpen
  - Imelda Ziekenhuis Bonheiden, Bonheiden, Mechelen
  - VITAZ, Sint-Niklaas, Oost-Vlaanderen
  - AZ Monica, Antwerp
  - Heilig Hartziekenhuis Lier, Lier
  - AZ Sint-Maarten, Mechelen

IPD SHARING:
Plan to Share IPD: No